CLINICAL TRIAL: NCT00894413
Title: A Phase II Trial of Tadalafil in Patients With Squamous Cell Carcinoma of the Upper Aero Digestive Tract
Brief Title: A Trial of Tadalafil in Patients With Squamous Cell Carcinoma of the Upper Aero Digestive Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: J0813; 1R21CA135635-01 (NIH); NA_00012749 (Other: JHM IRB)
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Pill
- Tadalafil (Experimental): Tadalafil 20 mg once per day
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — 20 mg once daily for 10 - 14 days
  Other Names: Cialis
  Arms: Tadalafil
Other: Placebo Pill — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this trial is to determine whether or not Cialis (tadalafil) administered to head and neck squamous cell cancer patients augments immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, previously untreated invasive head and neck squamous cell carcinoma OR histologically confirmed not yet treated recurrent head and neck squamous cell carcinoma (must be at least 3 months after diagnosis and completion of treatment for primary disease or last recurrence).
2. Disease location amenable to biopsy in outpatient clinical setting or operative biopsy within routine accepted schedule and practice of clinical care
3. No medical contraindication to biopsy of target lesion.
4. ECOG performance status 0-1
5. Required laboratory data (to be obtained within 4 weeks of initiation):

   * Platelets > 75,000/mm³
   * Calculated Creatinine Clearance (CRCL)> 60 mL/min iii. Total serum bilirubin < 1.5 mg/dL.
   * No intercurrent illness likely to prevent protocol therapy or surgical resection
6. Patients with a history of a curatively treated malignancy must be disease-free and have a survival prognosis that exceeds five years.
7. Female patients must not be pregnant or breast feeding. A negative pregnancy test is required within 14 days of randomization for all women of childbearing potential.
8. Willingness and ability to give signed written informed consent.

Exclusion Criteria:

1. Known severe hypersensitivity to tadalafil or any of the excipients of this product
2. Patients who have a concurrent malignancy or a history of previous malignancy treated with curative therapy within the last 3 months (other than squamous/basal cell cancer of the skin or cervical cancer) who have a survival prognosis of < 5 years.
3. Treatment with a non-approved or investigational drug within 30 days before day 1 of trial treatment.
4. Incomplete healing from previous oncologic or other major surgery.
5. Pregnancy or breast feeding (women of childbearing potential).
6. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
7. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial.
8. Current therapy with ketoconazole or oral antifungal therapy.
9. History of significant hypotensive episode requiring hospitalization.
10. A history of acute myocardial infarction within prior 3 months, uncontrolled angina,
11. Uncontrolled arrhythmia, or uncontrolled congestive heart failure
12. Age < 18
13. History of any of the following cardiac conditions:

    * Angina requiring treatment with long-acting nitrates.
    * Angina requiring treatment with short-acting nitrates within 90 days of planned tadalafil administration.
    * Unstable angina within 90 days of visit 1 (Braunwald 1989).
    * Positive cardiac stress test without documented evidence of subsequent, effective cardiac intervention.
14. History of any of the following coronary conditions within 90 days of planned tadalafil administration:

    * Myocardial Infarction.
    * Coronary artery bypass graft surgery.
    * Percutaneous coronary intervention (for example, angioplasty or stent placement).
    * Any evidence of heart disease (NYHA≥Class III as defined in Protocol Attachment LVHG.3) within 6 months of planned tadalafil administration
15. Current treatment with nitrates.
16. Current systemic treatment with a potent cytochrome P450 3A4 (CYP3A4) inhibitor such as ketoconazole or ritonavir.
17. Received treatment within the last 30 days with a drug or device that has not received regulatory approval for any indication at the time of Visit 1.
18. Prior chronic immune suppressive state (AIDS, immunosuppressive therapy).
19. History of hypotension and/or blindness during prior treatment with Tadalafil or other PDE-5 inhibitors.
20. prior history of non-arterial ischemic optic retinopathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-05-08 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Califano, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Result] Califano JA, Khan Z, Noonan KA, Rudraraju L, Zhang Z, Wang H, Goodman S, Gourin CG, Ha PK, Fakhry C, Saunders J, Levine M, Tang M, Neuner G, Richmon JD, Blanco R, Agrawal N, Koch WM, Marur S, Weed DT, Serafini P, Borrello I. Tadalafil augments tumor specific immunity in patients with head and neck squamous cell carcinoma. Clin Cancer Res. 2015 Jan 1;21(1):30-8. doi: 10.1158/1078-0432.CCR-14-1716. PMID 25564570

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects were screen failures
Period: Overall Study
Arm/Group | Placebo | Tadalafil
Started | 15 | 25
Completed | 15 | 17
Not Completed | 0 | 8
Not completed — Physician Decision | 0 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data was only collected in participants who completed study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (6) | 60 (15) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 13 | 16 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 14 | 27
  Black/other | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 17 | 32
Tobacco exposure [Count of Participants; unit: Participants] — Population: Data was not collected in 1/17 participants from tadalafil arm
  Participants
    Never: number analyzed (Participants) | 15 | 16 | 31
    Never | 8 | 2 | 10
    Ever: number analyzed (Participants) | 15 | 16 | 31
    Ever | 7 | 14 | 21
Ethanol (ETOH) Exposure [Count of Participants; unit: Participants] — Population: Data was not collected in 2/15 participants from the placebo arm and 3/17 participants from the tadalafil arm
  Participants
    Never: number analyzed (Participants) | 13 | 14 | 27
    Never | 6 | 4 | 10
    Ever: number analyzed (Participants) | 13 | 14 | 27
    Ever | 7 | 10 | 17
Site of Squamous Cell Carcinoma [Count of Participants; unit: Participants]
  Hypopharynx/larynx | 1 | 6 | 7
  Oral cavity | 5 | 2 | 7
  Oropharynx | 9 | 6 | 15
  Unknown | 0 | 3 | 3
Clinical stage [Count of Participants; unit: Participants] — Staging is defined by the American Joint Committee on Cancer (AJCC) TNM system where T= primary tumor, N= spread to nearby lymph nodes, Grade Group 1 through 4, and further letter staging. A lower number reflects less spread of cancer and a lower letter reflects a lower stage. Population: Data was not collected in 1/17 participants from tadalafil arm
  Participants
    Tumor (T) stage : T0/Tx/T1/T2: number analyzed (Participants) | 15 | 16 | 31
    Tumor (T) stage : T0/Tx/T1/T2 | 12 | 6 | 18
    Tumor (T) stage : T3/T4: number analyzed (Participants) | 15 | 16 | 31
    Tumor (T) stage : T3/T4 | 3 | 10 | 13
    Node (N) stage : N0/N1: number analyzed (Participants) | 15 | 16 | 31
    Node (N) stage : N0/N1 | 7 | 7 | 14
    Node (N) stage : N2/N3: number analyzed (Participants) | 15 | 16 | 31
    Node (N) stage : N2/N3 | 8 | 9 | 17
Human Papilloma Virus (HPV) status [Count of Participants; unit: Participants]
  Negative | 6 | 10 | 16
  Positive | 8 | 5 | 13
  Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Immune Response After Tadalafil Administration
Description: Median fold-change in immune response of T-cell expansion, delayed-type hypersensitivity reactions, CD4/CD69, CD8/CD69. A positive value indicates an increase in immune response.
Time Frame: Change from baseline to up to 14 days post-intervention
Population: Data was not evaluable in 1/15 participants from the placebo group, 2/17 participants in the tadalafil group (for T-cell expansion, CD4/CD69, CD/CD69) and 1/17 for DTH area.
Measure: Median (Full Range); unit: fold change
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 14 | 16
fold change
  T-cell expansion: number analyzed (Participants) | 14 | 15
  T-cell expansion | 1.13 [0.56 to 2.17] | 1.59 [0.73 to 6.31]
  DTH area | 1.14 [0.17 to 230] | 4.74 [0.27 to 80.0]
  CD4/CD69: number analyzed (Participants) | 14 | 15
  CD4/CD69 | 0.90 [0.44 to 3.10] | 1.29 [0.86 to 3.19]
  CD8/CD69: number analyzed (Participants) | 14 | 15
  CD8/CD69 | 0.93 [0.56 to 1.57] | 1.14 [0.94 to 2.88]

ADVERSE EVENTS:
Time Frame: up to 4 years
Arm/Group | Placebo | Tadalafil
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/25
Other Adverse Events (participants affected / at risk) | 0/15 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Tadalafil (N=25)
Chest Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — Pt started feeling chest tightness, he was evaluated in ER and admitted. Pt was evaluated for cardiac issues & a full cardiac workup was done. No cardiac problems were found was diagn as "acid reflux" and sent home with medication for acid reflux.
Fever (General disorders) | 1 (1) | 1 — Infection not related to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes